CLINICAL TRIAL: NCT05831540
Title: Clinical Decision Support Tools to Increase HPV Vaccination in Pharmacies
Brief Title: Clinical Decision Support Tools to Increase Human Papillomavirus (HPV) Vaccination in Adolescents in Pharmacies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study has been terminated due to the conclusion of funding. We were able to collect data on primary outcomes through pharmacy staff, but due to recruitment challenges were not able to complete secondary outcome recruitment.
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1122655; NCI-2023-01989 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11086 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-03-20; First posted 2023-04-26 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Human Papillomavirus-Related Carcinoma
MeSH Terms: interventions — Delivery of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (staff focus group) (Experimental): Staff participate in facilitated planning discussions to develop CDS tools on study.
  Interventions: Other: Discussion; Other: Survey Administration
- Group II (staff CDS tool utilization) (Experimental): Staff receives CDS tools training and implements CDS tools to facilitate HPV vaccination on study.
  Interventions: Other: Educational Activity; Behavioral: Healthcare Activity; Other: Survey Administration
- Group III (parent survey) (Experimental): Parents complete survey post-intervention on study.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Discussion — Participate in focus group
  Other Names: Discuss
  Arms: Group I (staff focus group)
Other: Educational Activity — Undergo training to use CDS tool
  Arms: Group II (staff CDS tool utilization)
Behavioral: Healthcare Activity — Utilize CDS tool
  Other Names: Health Care Activity; Healthcare
  Arms: Group II (staff CDS tool utilization)
Other: Survey Administration — Complete survey

SUMMARY:
This clinical trial develops and tests how well a clinical decision support (CDS) tool works to increase human papillomavirus (HPV) vaccination of children between the age of 9-17 (adolescents) in pharmacies. HPV vaccination rate in eligible adolescents remains low even though over 90% of the cancers in adults caused by HPV can be prevented by the HPV vaccine. The National Vaccine Advisory Committee recommends HPV vaccinations to be given in pharmacies to increase access to vaccines, but pharmacy processes and lack of awareness of the service among parents impact the use of local pharmacies for HPV vaccinations. Using a focus group may be an effective method to develop a CDS tool and create a process that may be more convenient for parents to get their adolescent's vaccine at their local pharmacy. A CDS tool may make it easier to obtain HPV vaccines, and as a result increase the adolescent HPV vaccination rate and reduce the incidence of cancer caused by HPV.

DETAILED DESCRIPTION:
OUTLINE: Participants are assigned to 1 of 3 groups.

Group I: Staff participate in facilitated planning discussions to develop CDS tools on study. (Aim I)

Group II: Staff receives CDS tools training and implements CDS tools to facilitate HPV vaccination on study. (Aim II)

Group III: Parents complete survey post-intervention on study. (Aim II)

ELIGIBILITY:
Inclusion Criteria:

* AIM I: >= 18 years
* AIM I: Pharmacy staff: Employed at the partnering community pharmacies in Washington state
* AIM I: Scientific Technologies Corportation (STC)Health staff: Employed at STCHealth
* AIM I: PioneerRx staff: Employed at PioneerRx
* AIM II: >= 18 years
* AIM II: Parents: English speaking parent or guardian of at least one child, ages 9-17, living in Washington state and obtained an HPV vaccination for their child at a participating pharmacy and have access to a telephone or computer with internet access.
* AIM II: Pharmacy staff: Employed at community pharmacies recruited into the study located in Washington state

Exclusion Criteria:

* Pharmacy staff: Floaters/per diem. Those who object to having the focus group discussions audio recorded. Those who object to participating in implementation evaluation surveys
* STCHealth staff: Those who object to having the focus group discussions audio recorded
* PioneerRx staff: Those who object to having the focus group discussions audio recorded
* Parents: Those who decline to provide feedback on their experiences with getting their children vaccinated at the pharmacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Development/refinement of the CDS tools to support and guide any adaptations to the pharmacy staff's vaccination workflow to improve vaccine delivery. (Aim 1) | Up to 6 months
  The research team will analyze the collected qualitative data using framework-guided rapid analyses described by Gale et al. The qualitative data will be used to direct and document the development and refinement process for the CDS tools to support HPV vaccination and to guide any adaptations to the pharmacy staff's vaccination workflow to improve their delivery of HPV vaccine. Adaptations made to a pharmacy's vaccination workflow will be methodically documented using Stirman's Taxonomy of Adaptation Characteristics.
Acceptability of CDS tools: Pharmacy staff (Aim II) | Post-implementation of CDS tools survey (at Months 11-12)
  Will use validated survey measure to assess pharmacy staff's report of the acceptability of the CDS tools to support HPV Vaccination.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Change in Acceptability of pharmacy-based HPV vaccination: Pharmacy staff (Aim II) | Pre-implementation of CDS Tools survey (at Months 4-5) and post- test implementation survey (at Months 11-12)
  The survey will ask pharmacy staff to respond to statements designed to measure acceptability of pharmacy-based HPV vaccination.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Acceptability of pharmacy-based HPV vaccination: Parents (Aim II) | Post-vaccination experience survey (at Months 8-12)
  The survey will ask parents to respond to statements designed to measure acceptability of their vaccine experience at the pharmacy.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Appropriateness of CDS tools: Pharmacy staff (Aim II) | Post-test implementation survey (at Months 11-12)
  The survey will ask pharmacy staff to respond to statements designed to measure appropriateness of the CDS tools to support HPV vaccination.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Appropriateness of pharmacy-based HPV vaccination: Pharmacy staff (Aim II) | Pre-test implementation survey (at Months 4-5) and post- test implementation survey (at Months 11-12)
  The survey will ask pharmacy staff to respond to statements designed to measure appropriateness of pharmacy-based HPV vaccination.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Appropriateness of pharmacy-based HPV vaccination: Parents (Aim II) | Post-vaccination experience survey (at Months 8-12)
  The survey will ask parents to respond to statements designed to measure appropriateness of their vaccine experience at the pharmacy.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Feasibility of CDS tools: Pharmacy staff (Aim II) | Post-test implementation survey (at Months 11-12)
  The survey will ask pharmacy staff to respond to statements designed to measure feasibility of the CDS tools to support HPV vaccination.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Feasibility of pharmacy-based HPV vaccination: Pharmacy staff (Aim II) | Pre-test implementation survey (at Months 4-5) and post- test implementation survey (at Months 11-12)
  The survey will ask pharmacy staff to respond to statements designed to measure feasibility of pharmacy-based HPV vaccination.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Feasibility of pharmacy-based HPV vaccination: Parents (Aim II) | Post-vaccination experience survey (at Months 8-12)
  The survey will ask parents to respond to statements designed to measure feasibility of their vaccine experience at the pharmacy.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Usability of CDS tools: Pharmacy staff (Aim II) | Post-test implementation survey (at Months 11-12)
  The survey will ask pharmacy staff to respond to statements designed to measure usability of the CDS tools to support HPV vaccination.
  Survey responses will include 5-point scales:
  1. = Not at all confident
  2. = Not very confident
  3. = Neither (neutral)
  4. = Moderately confident
  5. = Completely confident
  And
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
Parents' experience Survey (Aim II) | Post-implementation of CDS tools up to 12 months
  This is a 30-question survey asking about experience with getting child vaccinated at participating pharmacy.
  Survey responses will include a 5-point scales:
  1. = Strongly disagree
  2. = Somewhat disagree
  3. = Neither agree nor disagree
  4. = Somewhat agree
  5. = Strongly agree
  And
  1. Completely dissatisfied
  2. Somewhat dissatisfied
  3. Neither satisfied nor dissatisfied
  4. Somewhat satisfied
  5. Completely satisfied
HPV vaccination rate per pharmacist at each pharmacy (Aim II) | 12 months prior to CDS tool implementation (baseline) up to 5 months post-implementation
  Outcomes of implementation analyzed using nonparametric tests appropriate for small sample statistics, like Wilcoxon sign-rank test.

SECONDARY OUTCOMES:
Rate of other adolescent vaccinations per pharmacist at each pharmacy (Aim II) | 12 months prior to CDS tool implementation (baseline) up to 5 months post-implementation
  Outcomes of implementation analyzed using nonparametric tests appropriate for small sample statistics, like Wilcoxon sign-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT05831540/ICF_000.pdf